CLINICAL TRIAL: NCT00120198
Title: A Pilot Study of Cyclophosphamide/Pegylated Liposomal Doxorubicin/Vincristine/Prednisone (CDOP) Plus Rituximab for Treatment of Elderly Patients With Previously Untreated Non-Hodgkin's Lymphoma
Brief Title: Pegylated Liposomal Doxorubicin Containing Chemotherapy in the Treatment of Older Non-Hodgkin's Lymphoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Geriatric Oncology Consortium (Other)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOC-LY-010
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL; elderly
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

INTERVENTIONS:
Drug: CDOP plus rituximab

SUMMARY:
Currently there is no one standard of care for older patients with Non-Hodgkin's Lymphoma (NHL). The study will examine the tolerability and feasibility to the combination of Cyclophosphamide, Pegylated Liposomal Doxorubicin, Vincristine, Prednisone (CDOP) plus Rituximab.

DETAILED DESCRIPTION:
Elderly NHL patients tend to tolerate the combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) less well when compared to the younger population. Cardiotoxicity, as well as neutropenia, are the most common side effects in the elderly population with age being a risk factor for doxorubicin induced cardiac toxicity. Treatment related toxicity in the older population can preclude adequate therapy and potentially contribute to poor outcomes. Pegylated liposomal doxorubicin has shown similar efficacy with a significant lower incidence of cardiotoxicity ad significantly fewer cardiac events compared with conventional doxorubicin. Exploration of alternative regimens to maximize tolerability and thus enhance overall efficacy in this population is warranted. Both safety and efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older;
* Diagnosis of Non-Hodgkin's lymphoma where therapy with CHOP plus rituximab is considered;
* Previously untreated;
* ECOG 0-2
* Adequate renal and hepatic functions;
* Cardiac ejection fraction at least 50% by MUGA. No significant cardiac abnormalities by EKG;
* Signed informed consent

Exclusion Criteria:

* CNS involvement by lymphoma;
* Hypersensitivity to study drugs;
* Active infection;
* Prior treatment with monoclonal antibodies for cancer;
* History of cardiac disease with New York Heart Association Class II or greater or clinical evidence of congestive heart failure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and tolerability of CDOP plus rituximab in elderly patients with previously untreated NHL.

SECONDARY OUTCOMES:
Tumor response
duration of response
median time to disease progression
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lodovico Balducci, MD, Study Chair — Geriatric Oncology Consortium
Locations (5):
- United States (5):
  - Oxnard, California
  - Washington D.C., District of Columbia
  - Inverness, Florida
  - Lecanto, Florida
  - Belleville, New Jersey